CLINICAL TRIAL: NCT03085303
Title: Treatment of Atopic Dermatitis by a Full-Body Blue Light Device
Acronym: AD-Blue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland BV (Industry)
Collaborators: University Hospital Goettingen (Other); Philipps University Marburg (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FBB-CT01
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients are blinded by wearing tinted glasses for eye protection which disenable distinction of different wave lengths of light. Medical doctors will examine patients in other rooms than those equipped with the investigational medical devices. These examiners are blinded and are therefore not involved in the preparation and process of the irradiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blue light at 415nm (Experimental): Full body irradiation for 30min (15 min. each body side) with blue light at 415nm peak wavelength with full body blue device.
  Interventions: Device: Full Body Blue Light Device
- Blue light at 450nm (Experimental): Full body irradiation for 30min (15 min. each body side) with blue light at 450nm peak wavelength with full body blue device.
  Interventions: Device: Full Body Blue Light Device
- Placebo (Placebo Comparator): Full body irradiation for 30min (15 min. each body side) with blue light at 450nm peak wavelength with a low dose setting (not therapeutically active) of the full body blue device.
  Interventions: Device: Full Body Blue Light Device

INTERVENTIONS:
Device: Full Body Blue Light Device — Full body blue light irradiation (phototherapy) of atopic dermatitis patients.

SUMMARY:
Multicentric, placebo-controlled, double-blinded, three-armed, prospective, randomized controlled trial.150 patients diagnosed with atopic dermatitis will be randomized to arm 1 (irradiation for 30min at 415nm wavelength), arm 2 (irradiation for 30min at 450nm wavelength), and arm 3 (irradiation for 30min at low-dose (placebo)). Irradiation will be scheduled 3 times a week for 8 weeks. Patients will be followed up for four weeks after the last irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study mandated procedure
* Good health as determined by the Investigator
* Willing and able to comply with study requirements
* Atopic dermatitis (AD) fulfilling the United Kingdom (UK) criteria of AD
* Age between 18 and ≤ 75 years
* Reliable method of contraception for women of childbearing potential (i.e. low failure rate less than 1% per year; e.g. oral contraceptives, intrauterine device [IUD] or transdermal contraceptive patch)
* Willing to abstain from excessive sun / UV exposure (e.g. sunbathe, solarium) during the course of the study
* Body Mass Index ≥ 18 and ≤ 35

Exclusion Criteria:

General

* Inmates of psychiatric wards, prisons, or other state institutions
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Participation in another clinical trial within the last 30 days
* Pregnant or nursing women
* Risk of non-compliance with study procedures

Medical History

* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases may include cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease, and others.
* Clinically relevant abnormalities in hematology, or blood chemistry at screening.
* Positive HIV-1/2Ab, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCV-Ab) test at screening.
* Diastolic blood pressure above 95 mmHg.
* Febrile illness within 2 weeks prior to baseline visit.
* Alcohol or drug abuse within 12 months prior to screening (i.e., Regular daily consumption of more than 1 liter of beer or the equivalent quantity of approximately 40 g of alcohol in another form.)
* Photodermatosis and/or significant photosensitivity, including porphyria and/or hypersensitivity to porphyrins as well as photosensitivity due to present or past (within the last year) intake of amiodarone.
* Congenital or acquired immunodeficiency
* Patients who have been diagnosed with invasive skin cancer at any time (=malignant cells invaded below the basal membrane of the epidermis), or with severe actinic damage present at baseline visit.
* Patients with genetic deficiencies attached with increased sensitivity to light or increased risk to dermatologic cancer (i.e. Xeroderma pigmentosum, Cockayne Syndrome, Bloom-Syndrome).

Concomitant medication/treatment in medical history and during the study

Within 8 weeks prior to baseline visit:

* Systemic immunosuppression treatment (steroids, cyclosporine, azathioprine, Mycophenolate Mofetil (MMF))

Within 4 weeks prior to baseline visit:

* UV radiation treatment

Within 2 weeks prior to baseline visit:

* Topical steroid treatment
* Topical calcineurin inhibitor treatment

Within 3 days prior to baseline visit:

* Photo-sensitising medication (e.g. psoralen, tetracyclines, hydrochlorothiazide, phenothiazines, quinolones, hypericumperforatum, arnica, valerian, tar) as assessed by the regular medication plan of the patient
* colours (e.g. thiazide, toluidine blue, eosin, methylene blue, rose Bengal, acridine) which will be visible on the patient's skin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Eczema Area Severity Index (EASI) at end of treatment | week 8
  Change in EASI from baseline to week 8

SECONDARY OUTCOMES:
Change in Score of Atopic Dermatitis (SCORAD) at end of treatment | week 8
  Change in SCORAD from baseline to week 8
Change in Patient Oriented Score of Atopic Dermatitis (PO-SCORAD) at end of treatment | week 8
  Change in PO-SCORAD from baseline to week 8
Change in Investigator Global assessment (IGA)at end of treatment | week 8
  Change in IGA from baseline to week 8
Change in itch Visual Analogue Scale (VAS) at end of treatment | week 8
  Change in itch VAS from baseline to week 8
EASI 50% | week 8
  Proportion of patients achieving 50% reduction from baseline EASI score at end of treatment
Change in Dermatology Life Quality Index (DLQI) at end of treatment | week 8
  Change in DLQI from baseline to week 8
Change in EASI at follow-up | week 12
  Change in EASI from end of treatment to week 12
Time until treatment response | week 0-8
  Time until Treatment Response is seen

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schoen, Prof, Principal Investigator — University Medical Center Göttingen, Clinic of Dermatology, Venereology and Allergology
Locations (3):
- Germany (2):
  - University Hospital Goettingen, Göttingen
  - University Hospital Marburg, Marburg
- University Hospital Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keemss K, Pfaff SC, Born M, Liebmann J, Merk HF, von Felbert V. Prospective, Randomized Study on the Efficacy and Safety of Local UV-Free Blue Light Treatment of Eczema. Dermatology. 2016;232(4):496-502. doi: 10.1159/000448000. Epub 2016 Aug 19. PMID 27537360
- [Derived] Buhl T, Santibanez Santana M, Forkel S, Kromer C, Seidel J, Mobs C, Pfutzner W, Pfeiffer S, Laubach HJ, Boehncke WH, Liebmann J, Born M, Schon MP. Full-body blue light irradiation as treatment for atopic dermatitis: a randomized sham-controlled clinical trial (AD-Blue). J Dtsch Dermatol Ges. 2023 Dec;21(12):1500-1510. doi: 10.1111/ddg.15211. Epub 2023 Oct 9. PMID 37814388
- [Derived] Kromer C, Nuhnen VP, Pfutzner W, Pfeiffer S, Laubach HJ, Boehncke WH, Liebmann J, Born M, Schon MP, Buhl T. Treatment of Atopic Dermatitis Using a Full-Body Blue Light Device (AD-Blue): Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 8;8(1):e11911. doi: 10.2196/11911. PMID 30622089